CLINICAL TRIAL: NCT04907552
Title: Forensic Dental Age Estimation : Validation of Computed Tomography for Third Mandibular Molar Demirjian's Staging Method in a 0- 25 Years French Living Population
Brief Title: Forensic Dental Age Estimation : Validation of Computed Tomography for Third Molar Demirjian's Staging
Acronym: SCAO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0576
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Mandible Fracture
Keywords: Dental age estimation; CT scan; dental panoramic; Validation CT scan; Radiography
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Age can be estimated in different ways by using skeletal age and dental age. Currently, bone age is determine thanks to the wrist x-rayed, and the dental age using variation in mineralization (Demirjian's score) on the dental panoramic (Mincer 1993).

More recently, reviews indicate the Computed tomography (CT) scan of the medial clavicular epiphysics can contribute to improve the accuracy of individual's age estimation (Houpert, 2016).

Furthermore, with the recent advances, the very low dose CT scan acquisitions can be perform with sufficient quality for the teeth analysis.

The goal of this study is to validate the use of dental CT for Demirjdian's staging method.

ELIGIBILITY:
Inclusion criteria:

* Patient aged between 0 and 25 years old
* Complete dental panoramic
* CT scan including mandible and maxilla
* Maximum of 2 months between CT scan and dental panoramic
* Medical imaging available on the PACS

Exclusion criteria:

* Medical imaging missing on the PACS
* Patient refuses to participate

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient aged between 0 and 25 years old
Sampling Method: Probability Sample
Enrollment: 557 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
weighted Kappa test between CT scan | day 1
  weighted Kappa test between CT scan and dental panoramic assessment of Demirjian's staging of third mandibular molar

SECONDARY OUTCOMES:
Mineralization difference | day 1
  Mineralization difference between mandibular and maxillar third molar
Dental age estimation in a south french population | day 1
  Dental age estimation in a south french population

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CYTEVAL, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC